CLINICAL TRIAL: NCT04510857
Title: Motivating Occupational Virtual Experiences In Therapy for Kids (MOVE-IT)
Brief Title: Motivating Occupational Virtual Experiences In Therapy for Kids
Acronym: MOVE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barron Associates, Inc. (Industry)
Collaborators: University of Virginia (Other); Duke University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOVE-IT; 5R44HD092169-03 (NIH)
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Virtual Reality; Occupational Therapy
Keywords: Cerebral palsy; Occupational therapy; Virtual reality; Therapy games; Pediatric hemiplegia; Teletherapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Intervention group performs home exercise program using the computer-aided MOVE-IT system for upper extremity therapy.
  Control group participants will be followed as they continue to receive their previously prescribed therapy services.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator administrating assessments will be blinded to subject group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- MOVE-IT Home Exercise Program (HEP) (Experimental): Participants will be asked to employ the MOVE-IT system for upper extremity practice at home 1 hour/day, 5 days/week over a 10-week period.
  Interventions: Device: MOVE-IT Intervention
- Usual Care Treatment (UCT) Control (Active Comparator): Children in the UCT group will be followed as they continue to receive their previously prescribed therapy services. These children will not receive any treatment services through the study as UCT group participants.
  Interventions: Behavioral: UCT Control

INTERVENTIONS:
Device: MOVE-IT Intervention — The MOVE-IT device comprises a custom smart toy and therapy game software to enable repetitive task practice involving the arm and hand.
  Arms: MOVE-IT Home Exercise Program (HEP)
Behavioral: UCT Control — Participants assigned to the UCT control group will continue to receive their previously prescribed therapy services.
  Arms: Usual Care Treatment (UCT) Control

SUMMARY:
A rater-blinded randomized controlled trial (RCT) will be conducted to compare the efficacy of MOVE-IT use in a remotely supervised home exercise program (HEP) to usual care for recovery of upper extremity (UE) function in children with hemiplegia.

DETAILED DESCRIPTION:
A rater-blinded randomized controlled trial (RCT) will be conducted to compare the efficacy of MOVE-IT use in a remotely supervised home exercise program (HEP) to usual care for recovery of upper extremity (UE) function in children with hemiplegia, and to acquire evidence of usability and acceptance of the MOVE-IT system by children and parents. The University of Virginia (UVA) will serve as coordinating center and single IRB for the two-site RCT that includes UVA and Duke University.

The primary Phase II investigational objective is to show a differential effect on the pre- to post-intervention change in UE motor function between an interventional group receiving the MOVE-IT HEP and a usual care treatment (UCT) group, as assessed by the Jebsen Tailor Hand Function Test (JTHFT), a time-based measure of functional hand motor skills, and other gold-standard clinical instruments for UE function including the Quality of Upper Extremity Skills Test (QUEST), with qualitative assessment of discrete movements, and the Wolf Motor Function Test (WMFT), which includes both quantitative and qualitative assessment of functional movements.

The pre-to-post intervention change in the composite JTHFT score will be the primary endpoint for the Phase II efficacy study. Secondary analysis will include pre-to-post intervention changes in the composite QUEST and WMFT scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemiplegia resulting from cerebral palsy, stroke, or other form of brain injury;
* Medically stable;
* Participant has antigravity strength in the affected UE at the elbow to at least 45 degrees of active flexion;
* Participant has antigravity shoulder strength in the affected UE to at least 30 degrees each in active flexion, abduction/adduction, and 15 degrees in active internal/external rotation when in an upright and seated position;
* Participant has ability to perform a basic color-matching test and identify characters on a vision chart;
* Participant must be available to attend study visits during an approximately 3-week participation period;
* Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

* History of uncontrolled seizures;
* Has received another form of intensive UE therapy, such as CIMT, within the prior 6 months;
* Unwillingness or inability to understand or follow verbal directions;
* Diagnosis of moderate to severe cortical-visual impairment that in the judgement of the Principal Investigator could adversely impact the subject's participation;
* Psychological diagnosis that in the determination of the Principal Investigator could significantly impact subject's participation or that could be aggravated by study participation;
* Determination that participation would result in over exertion, or significant discomfort or pain;
* Determination that participation would result in significant agitation or elevated stress;
* Visual field deficit in either eye that impairs the ability to view the computer monitor.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of Virginia (UVA), Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only children were considered enrolled in the study. A parent or legal guardian provided permission and the child verbal assented.
  Of the subjects enrolled, 2 failed screening tests (described in the protocol) and 2 others dropped out prior to randomization due to medical or personal reasons.
Period: Overall Study
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Started | 11 | 10
Completed | 10 | 8
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Analysis is for subjects enrolled and randomized to a treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Median (Full Range); unit: years] | 9 [6 to 12] | 6.5 [4 to 12] | 8.5 [4 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Pre Jebsen Taylor Hand Function Test (JTHFT)
Description: The JTHFT assesses hand function through timed movements such as simulated page turning, eating, stacking objects, and lifting objects of different size and mass. The JTHFT total score is simply the sum of all timed movements (in seconds). A lower score represents a better outcome.
Time Frame: Pre-intervention at Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 8
seconds | 433.9 (225.1) | 294.7 (217.3)

2. Primary Outcome: Post Jebsen Taylor Hand Function Test (JTHFT)
Description: as for outcome 1
Time Frame: Post Intervention at 10 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 8
seconds | 416.6 (228.9) | 268.3 (212.4)

3. Secondary Outcome: Pre Pediatric Motor Activity Log (Amount)
Description: The Pediatric Motor Activity Log (Amount) is a parent-reported assessment tool designed to evaluate the frequency of use of a child's affected (weaker) upper limb during 22 specific daily activities, such as reaching, grasping, or manipulating objects. For each activity, parents rate how often the child uses their affected arm on a 6-point Likert scale, ranging from 0 to 5. A score of 0 indicates that the child never uses the weaker arm for the activity (or the activity is not performed), while a score of 5 indicates that the weaker arm is used as frequently as the stronger arm for that activity. The reported score is the average of the individual scores for the 22 activities. A higher score represents a better outcome.
Time Frame: Pre-intervention at Baseline
Population: PMAL data were missing for one UCT subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 7
score on a scale | 1.68 (0.60) | 2.30 (0.93)

4. Secondary Outcome: Post Pediatric Motor Activity Log (Amount)
Description: as for outcome 3
Time Frame: Post Intervention at 10 weeks
Population: PMAL data were missing for one UCT subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 7
score on a scale | 1.80 (0.73) | 2.23 (0.93)

5. Secondary Outcome: Pre Pediatric Motor Activity Log (How Well)
Description: The Preschool Pediatric Motor Activity Log (PMAL-How Well) is a parent-reported assessment tool designed to evaluate the quality of use of a child's affected upper limb (weaker arm) during 22 specific daily activities. For each activity, the parent rates the quality of their child's performance using the affected arm on a 6-point Likert scale, ranging from 0 to 5. A score of 0 indicates that the child does not use the weaker arm at all for the activity (or the activity is not performed), while a score of 5 indicates that the weaker arm is used as effectively as the stronger arm, with normal or near-normal quality of movement. The reported score is the average of the individual scores for the 22 activities. A higher score represents a better outcome.
Time Frame: Pre-intervention at Baseline
Population: PMAL data were missing for one UCT subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 7
score on a scale | 1.68 (0.95) | 2.73 (0.88)

6. Secondary Outcome: Post Pediatric Motor Activity Log (How Well)
Description: as for outcome 5
Time Frame: Post Intervention at 10 weeks
Population: PMAL data were missing for one UCT subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 7
score on a scale | 2.25 (0.73) | 2.98 (0.66)

7. Secondary Outcome: Pre Intervention Wolf Motor Function Test Time (WMFT-TIME)
Description: The WMFT test is a functionally-oriented clinical and research instrument. The test consists of 15 motor tasks scored both for time and quality of movement. WMFT-TIME is a quantitative measure calculated using the average time to complete the tasks. Any time greater than 120 seconds is recorded as 120 seconds. A patient's WMFT-TIME score (average completion time) thus ranges from 0 to 120. A reduction in WMFT-TIME implies improved motor function.
Time Frame: Pre-intervention at Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 8
seconds | 24.3 (17.2) | 18.3 (25.1)

8. Secondary Outcome: Post Intervention Wolf Motor Function Test Time (WMFT-TIME)
Description: as for outcome 7
Time Frame: Post Intervention at 10 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 8
seconds | 24.1 (18.7) | 24.9 (40.0)

9. Secondary Outcome: Pre Intervention Wolf Motor Function Test Functional Assessment (WMFT-FA)
Description: The WMFT test is a functionally-oriented clinical and research instrument. The test consists of 15 motor tasks scored both for time and quality of movement.
  The WMFT Functional Assessment (WMFT-FA) score is an observational assessment of movement quality and scored using a 6-point ordinal rating scale that ranges from 0 (no use of the affected side attempted) to 5 (normal function). A total WMFT-FA score is calculated by taking the average across all 15 UE tasks. A patient's WMFT-FA score is thus a real number that can range from 0 to 5. An increase in WMFT-FA score implies improved motor function.
Time Frame: Pre-intervention at Baseline
Population: WMFT FA data were missing for one UCT subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 7
score on a scale | 2.95 (0.92) | 3.40 (0.79)

10. Secondary Outcome: Post Intervention Wolf Motor Function Test Functional Assessment (WMFT-FA)
Description: as for outcome 9
Time Frame: Post Intervention at 10 weeks
Population: WMFT FA data were missing for one UCT subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 10 | 7
score on a scale | 3.00 (0.83) | 3.63 (0.74)

11. Secondary Outcome: Pre Quality of Upper Extremity Skills Test (QUEST)
Description: Quality of Upper Extremity Skills Test (QUEST) is a standardized assessment tool designed to evaluate upper extremity (UE) function in children with neuromotor disabilities, such as cerebral palsy. This study used only the dissociated movements and grasp function components of the QUEST instrument. Observational criteria were used to assign a value of 0, 1, or 2 for each of 44 items. Individual component scores were summed to create a total score with a range from 0 to 88. A higher value corresponds to a better outcome.
Time Frame: Pre-intervention at Baseline
Population: QUEST data were missing for 2 HEP subjects and 1 UCT subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 8 | 7
score on a scale | 67.5 (9.7) | 77.7 (8.5)

12. Secondary Outcome: Post Quality of Upper Extremity Skills Test (QUEST)
Description: as for outcome 11
Time Frame: Post Intervention at 10 weeks
Population: QUEST data were missing for 2 HEP subjects and 1 UCT subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
Number analyzed (Participants) | 8 | 7
score on a scale | 65.3 (9.7) | 77.4 (10.8)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | MOVE-IT Home Exercise Program (HEP) | Usual Care Treatment (UCT) Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04510857/Prot_SAP_000.pdf